CLINICAL TRIAL: NCT00121108
Title: A Phase 3 Study of MEDI-524 (Motavizumab), an Enhanced Potency Humanized Respiratory Syncytial Virus (RSV) Monoclonal Antibody, for the Prevention of RSV Disease Among Native American Infants in the Southwestern United States
Brief Title: MEDI-524 (Motavizumab) for the Prevention of Respiratory Sycytial Virus (RSV) Disease Among Native American Indian Infants in the Southwestern United States
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP117
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Healthy
Keywords: RSV, infants, Native American Indians
MeSH Terms: interventions — motavizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive IM dose of placebo matched to motavizumab every 30 days for a maximum of 5 injections (on Days 0, 30, 60, 90, and 120) during the the RSV season.
  Interventions: Other: Placebo
- Motavizumab (Active Comparator): Participants will receive IM dose of motavizumab 15 milligram/Kilogram (mg/kg) every 30 Days for a maximum of 5 injections (on Days 0, 30, 60, 90, and 120) during the RSV season.
  Interventions: Biological: Motavizumab

INTERVENTIONS:
Biological: Motavizumab — Intramuscular dose of motavizumab 15 mg/kg will be administered every 30 Days for a maximum of 5 injections (on Days 0, 30, 60, 90, and 120) during the RSV season.
  Other Names: MEDI-524
  Arms: Motavizumab
Other: Placebo — Intramuscular dose of placebo matched to motavizumab will be administered every 30 days for a maximum of 5 injections (on Days 0, 30, 60, 90, and 120) during the the RSV season.
  Arms: Placebo

SUMMARY:
MI-CP117 was a Phase 3, randomized, double-blind, placebo-controlled trial designed to determine if motavizumab is more effective than placebo in reducing RSV hospitalization in otherwise healthy Native American Infants in the Southwestern United States during their first RSV season.

DETAILED DESCRIPTION:
MI-CP117 was a Phase 3, randomized, double-blind, placebo-controlled trial designed to determine if motavizumab is more effective than placebo in reducing RSV hospitalization in otherwise healthy Native American infants during their first RSV season.

Participants were randomized in a 2:1 ratio to receive either 15 mg/kg motavizumab or placebo by intramuscular (IM) injection every 30 days during the RSV season for a maximum of 5 injections.

During their first RSV season, participants were evaluated monthly just prior to each injection of study drug for adverse events (AEs) (including medically attended otitis media), with a final post-dosing follow up evaluation at Study Day 150. During Seasons 1, 2, and 3, blood was to be collected prior to the first and last dose of study drug for serum chemistry evaluations, motavizumab serum concentrations, and anti-motavizumab antibodies. Efficacy and safety outcomes were examined through Study Day 150 and wheezing outcomes were evaluated from the time of randomization until the third birthday.

ELIGIBILITY:
Inclusion Criteria:

* 6 months of age or younger at randomization (child must be randomized on or before their 6-month birthday)
* Male or female Native American
* General state of good health
* Written informed consent obtained from the participant's parent(s) or legal guardian

Exclusion Criteria:

* Gestational age less than or equal to 35 weeks
* Chronic lung disease of prematurity
* A bleeding diathesis that would preclude IM injections
* Hospitalization at the time of randomization (unless discharge is anticipated within 10 days)
* Active RSV infection (a child with signs/symptoms of respiratory infection must have negative RSV testing) or known prior history of RSV infection
* A documented wheezing episode before enrollment
* Known renal impairment
* Known hepatic dysfunction
* Clinically significant congenital anomaly of the respiratory tract
* Chronic seizure or evolving or unstable neurologic disorder
* Congenital heart disease (CHD) (children with uncomplicated CHD [e.g., Patent ductus arteriosus, small septal defect] and children with complicated CHD who are currently anatomically and hemodynamically)
* Known immunodeficiency
* Mother with human immunodeficiency virus infection (unless the child has been proven to be not infected)
* Known allergy to Ig products
* Receipt of palivizumab, Respiratory syncytial virus immunoglobulin, intravenous (RSV-IGIV), or other RSV-specific monoclonal antibody, or any other polyclonal antibody (for example, hepatitis B immunoglobulin, IVIG) within 3 months prior to randomization
* Anticipated use of palivizumab or IVIG during the study (blood transfusions permitted)
* Previous receipt of RSV vaccines
* Participation in other investigational drug product studies
* Any medical or social condition which, in the opinion of the investigator, would adversely affect monitoring the infant
* Inability to complete the study follow-up period through up to 5 years of age

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2127 (Actual)
Dates: Start 2004-11-15 (Actual); Primary Completion 2010-12-27 (Actual); Study Completion 2010-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune, LLC MedImmune, LLC, Study Director — MedImmune LLC
Locations (12):
- United States (12):
  - Research Site, Chinle, Arizona
  - Research Site, Cibecue, Arizona
  - Research Site, Fort Definace, Arizona
  - Research Site, San Carlos, Arizona
  - Research Site, Tuba City, Arizona
  - Research Site, Whiteriver, Arizona
  - Research Site, Winslow, Arizona
  - Research Site, Baltimore, Maryland
  - Research Site, Bloomfield, New Mexico
  - Research Site, Crownpoint, New Mexico
  - Research Site, Gallup, New Mexico
  - Research Site, Shiprock, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] O'Brien KL, Chandran A, Weatherholtz R, Jafri HS, Griffin MP, Bellamy T, Millar EV, Jensen KM, Harris BS, Reid R, Moulton LH, Losonsky GA, Karron RA, Santosham M; Respiratory Syncytial Virus (RSV) Prevention study group. Efficacy of motavizumab for the prevention of respiratory syncytial virus disease in healthy Native American infants: a phase 3 randomised double-blind placebo-controlled trial. Lancet Infect Dis. 2015 Dec;15(12):1398-408. doi: 10.1016/S1473-3099(15)00247-9. Epub 2015 Nov 4. PMID 26511956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 15 Nov 2004 to 27 Dec 2010 in the United States of America.
Groups:
- Placebo: Participants received intramuscular (IM) dose of placebo matched to motavizumab every 30 days for a maximum of 5 injections (on Days 0, 30, 60, 90, and 120) during the respiratory syncytial virus (RSV) season.
- Motavizumab: Participants received IM dose of motavizumab 15 milligram/Kilogram (mg/kg) every 30 Days for a maximum of 5 injections (on Days 0, 30, 60, 90, and 120) during the RSV season.
Period: Overall Study
Arm/Group | Placebo | Motavizumab
Started | 710 | 1417
Completed | 589 | 1192
Not Completed | 121 | 225
Not completed — Lost to Follow-up | 10 | 22
Not completed — Withdrawal by Subject | 106 | 195
Not completed — Death | 5 | 8

BASELINE CHARACTERISTICS:
Population: The Intent to treat (ITT) population included all participants in the treatment group according to their randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Motavizumab | Total
Number analyzed (Participants) | 710 | 1417 | 2127
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.13 (1.89) | 2.08 (1.92) | 2.10 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 343 | 710 | 1053
  Male | 367 | 707 | 1074
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Navajo | 576 | 1149 | 1725
  White Mountain Apache | 102 | 203 | 305
  San Carlos Apache | 15 | 28 | 43
  Zuni | 0 | 1 | 1
  Hopi | 8 | 19 | 27
  Other - Not specified | 9 | 17 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Syncytial Virus (RSV) Hospitalization
Description: An RSV hospitalization is defined as either 1) a respiratory hospitalization with a positive central real-time reverse transcription polymerase chain reaction (RT-PCR) RSV test collected within 3 days of hospitalization or 2) new onset of lower respiratory symptoms in an already hospitalized child, with an objective measure of worsening respiratory status and positive RSV test.
Time Frame: From study Day 0 through study Day 150
Population: The ITT population included all participants in the treatment group according to their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 710 | 1417
Participants | 80 | 21
Statistical Analysis 1: Comparison: Placebo vs Motavizumab; Test type: Superiority; p < 0.001, Fisher Exact; Relative risk = 0.13, 95% CI 2-sided [0.08 to 0.21]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From study Day 0 through study Day 150
Population: Safety population included all the participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 708 | 1414
Participants
  TEAEs | 686 | 1361
  TESAEs | 148 | 212

3. Secondary Outcome: Number of Participants With RSV Outpatient Medically Attended Lower Respiratory Illness (MA LRI)
Description: The RSV outpatient MA LRI was defined as an outpatient medically attended event designated as a lower respiratory illness with a positive RT-PCR RSV test. An LRI event is one that has a medical diagnosis of bronchiolitis or pneumonia. In the absence of such a medical diagnosis, the occurrence of LRI events was determined by the principal investigator after review of the medical record and considering the presence of cough, retractions, rhonchi, wheezing, crackles, or rales, associated with symptoms (by history or clinical findings) of coryza, fever, or apnoea.
Time Frame: From study Day 0 through study Day 150
Population: The ITT population included all participants in the treatment group according to their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 710 | 1417
Participants | 71 | 41

4. Secondary Outcome: Number of Participants With Medically Attended-Otitis Media (MA-OM) Events
Description: Otitis media (OM) was recorded as the diagnosis if the following terms were used by the medical care provider: acute OM, acute tympanic membrane (TM) perforation, bulging TM, red TM with fever, OM with effusion, or middle ear effusion. A new episode was defined as a physician-diagnosed OM in either ear after a normal middle ear exam of the ear in question or an episode of acute OM greater than or equal to 21 days after resolution of the previous episode. A diagnosis of persistent middle ear effusion was not recorded as a new OM event.
Time Frame: From study Day 0 through study Day 150
Population: The ITT population included all participants in the treatment group according to their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 710 | 1417
Participants | 275 | 532

5. Secondary Outcome: Number of Participants With Frequency of MA-OM Events
Description: Otitis media was recorded as the diagnosis if the following terms were used by the medical care provider: acute OM, acute TM perforation, bulging TM, red TM with fever, OM with effusion, or middle ear effusion. A new episode was defined as a physician-diagnosed OM in either ear after a normal middle ear exam of the ear in question or an episode of acute OM greater than or equal to 21 days after resolution of the previous episode. A diagnosis of persistent middle ear effusion was not recorded as a new OM event. Number of participants with frequency of MA-OM events (either 0, 1, 2, 3, or greater than [>] 3) are reported.
Time Frame: From study Day 0 through study Day 150
Population: The ITT population included all participants in the treatment group according to their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 710 | 1417
Participants
  MA OM: 0 | 435 | 885
  MA OM: 1 | 190 | 372
  MA OM: 2 | 55 | 114
  MA OM: 3 | 26 | 32
  MA OM: >3 | 4 | 14

6. Secondary Outcome: Number of Participants With Medically Attended Wheezing Episodes
Description: Wheezing events were included in the analysis of medically-attended wheezing, if the medical care provider documented wheezing in the medical record or records as a discharge diagnosis any of asthma, bronchiolitis, wheezing, or reactive airway disease. A new wheezing episode was recorded as one that occurred >2 weeks after the diagnosis of the previous episode and the medical opinion was that the wheezing does not represent a persistence of the previous episode. Number of participants with greater than or equal to (>=) 1 MA wheezing events and >= 3 MA wheezing events occurring from first through 3 years of age are reported.
Time Frame: From first year through 3 years
Population: The ITT population included all participants in the treatment group according to their randomized treatment group. Here, "number analyzed" signified, only those participants who were analyzed from first year through 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 641 | 1278
Participants
  >= 1 MA wheezing events | 179 | 342
  >= 3 MA wheezing events | 16 | 35

7. Secondary Outcome: Number of Participants With Serious Early Childhood Wheezing Episodes
Description: Serious early childhood wheezing (SECW) was defined as: three or more medically attended wheezing events over a 12 month period occurring any time from the first through the third birthday, or a need for one or more courses of systemic steroids for a treatment of a medically attended wheezing event from the first through the third birthday, or a need for asthma-controller medication over a 12 month period for at least 3 consecutive months (>= 90 days) or 5 cumulative months (>= 150 days) any time from the first through the third birthday, or at least one inpatient wheezing event from the first through the third birthday.
Time Frame: From first year through 3 years
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 641 | 1278
Participants
  SECW | 90 | 190
  Three or more MA wheezing events over a 12 month period | 16 | 35
  Need of systemic steroids for a MA wheezing event | 66 | 144
  Asthma-controller medication for wheezing over a 12 month period | 2 | 11
  >= 1 hospitalization with MA wheezing | 47 | 91

8. Secondary Outcome: Number of Participants With Frequency of Medically Attended Wheezing Events
Description: Wheezing events were included in the analysis of medically-attended wheezing, if the medical care provider documented wheezing in the medical record or records as a discharge diagnosis any of asthma, bronchiolitis, wheezing, or reactive airway disease. A new wheezing episode was recorded as one that occurred >2 weeks after the diagnosis of the previous episode and the medical opinion is that the wheezing does not represent a persistence of the previous episode. Number of participants with frequency of MA wheezing events (either 0, 1, 2, 3, 4, or greater than or equal to [>=] 5) are reported.
Time Frame: Study Day 0 through 3 years
Population: The ITT population included all participants in the treatment group according to their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab
Number analyzed (Participants) | 710 | 1417
Participants
  0 events | 384 | 908
  1 event | 182 | 288
  2 events | 72 | 109
  3 events | 34 | 44
  4 events | 18 | 27
  >= 5 events | 20 | 41

9. Secondary Outcome: Mean Trough Serum Concentrations of Motavizumab
Description: The mean trough serum concentrations of motavizumab are reported.
Time Frame: Day 0 (pre Dose 1) and Day 120 (Pre Dose 5)
Population: Pharmacokinetics (PK) population included all participants (in seasons 1 through 3) who received at least 4 doses of motavizumab and had a post-baseline PK measurement available. Here, number analyzed signified only those participants who had adequate PK samples at the specified time points.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Motavizumab
Number analyzed (Participants) | 509
μg/mL
  Day 0 (Pre dose 1): number analyzed (Participants) | 495
  Day 0 (Pre dose 1) | 0.003212 (0.07147)
  Day 120 (pre dose 5) | 86.46 (31.77)

10. Secondary Outcome: Number of Participants With Positive Anti-Motavizumab Antibodies After Full Dose
Description: The number of participants with positive serum antidrug antibodies (ADAs) to motavizumab after full dose are reported.
Time Frame: Day 0 (Pre Dose 1) and Day 120 (Pre Dose 5)
Population: Evaluable population for full dose included all participants (in season 1 through 3) who received 4 doses of motavizumab prior to ADA sample collection, and had Day 120 ADA data available. Here, number analyzed signified only those participants who had adequate ADA samples at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Motavizumab
Number analyzed (Participants) | 665
Participants
  Day 0 (Pre Dose 1): number analyzed (Participants) | 5
  Day 0 (Pre Dose 1) | 0
  Day 120 (Pre Dose 5) | 3

11. Secondary Outcome: Number of Participants With Positive Anti-Motavizumab Antibodies After Any Dose
Description: The number of participants with positive serum ADA to motavizumab after any dose are reported.
Time Frame: Day 0 (Pre Dose 1) and Day 120 (Pre Dose 5)
Population: Evaluable population for any dose included all participants (in season 1 through 3) who received at least 1 dose of motavizumab prior to ADA sample collection, and had Day 120 ADA data available. Here, number analyzed signified only those participants who had adequate ADA samples at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Motavizumab
Number analyzed (Participants) | 717
Participants
  Day 0 (Pre Dose 1): number analyzed (Participants) | 5
  Day 0 (Pre Dose 1) | 0
  Day 120 (Pre Dose 5) | 3

ADVERSE EVENTS:
Time Frame: From study Day 0 through study Day 150
Description: Safety population included all the participants who received any study drug.
Arm/Group | PLACEBO | MOTAVIZUMAB
All-Cause Mortality (participants affected / at risk) | 5/708 | 8/1414
Serious Adverse Events (participants affected / at risk) | 148/708 | 212/1414
Other Adverse Events (participants affected / at risk) | 682/708 | 1345/1414
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=708) | MOTAVIZUMAB (N=1414)
Benign familial neonatal convulsions (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Combined immunodeficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Fallot's tetralogy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Microvillous inclusion disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever neonatal (General disorders) | 4 (4) | 10 (11)
Pyrexia (General disorders) | 3 (3) | 8 (8)
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 (6) | 10 (11)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 4 (4)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 3 (3) | 3 (3)
Bronchiolitis (Infections and infestations) | 35 (36) | 29 (32)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Croup infectious (Infections and infestations) | 1 (1) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 14 (14) | 31 (32)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 5 (5)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 3 (3) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 8 (9)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Meningitis candida (Infections and infestations) | 0 (0) | 1 (1)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 20 (21) | 36 (39)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 6 (6) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 4 (4)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 38 (39) | 16 (17)
Respiratory syncytial virus infection (Infections and infestations) | 4 (5) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 6 (6) | 5 (5)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Bacterial test (Investigations) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 1 (1) | 0 (0)
Laboratory test interference (Investigations) | 1 (1) | 0 (0)
Medical observation (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Craniosynostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 5 (5)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Victim of child abuse (Social circumstances) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=708) | MOTAVIZUMAB (N=1414)
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 4 (4) | 23 (24)
Cerumen impaction (Ear and labyrinth disorders) | 39 (40) | 81 (94)
Ear pain (Ear and labyrinth disorders) | 8 (8) | 24 (24)
Conjunctivitis (Eye disorders) | 136 (152) | 271 (303)
Eye discharge (Eye disorders) | 12 (12) | 21 (21)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 26 (26)
Constipation (Gastrointestinal disorders) | 57 (61) | 97 (107)
Diarrhoea (Gastrointestinal disorders) | 106 (130) | 196 (230)
Enteritis (Gastrointestinal disorders) | 4 (4) | 17 (17)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 (10) | 19 (19)
Teething (Gastrointestinal disorders) | 86 (96) | 167 (178)
Vomiting (Gastrointestinal disorders) | 22 (23) | 49 (50)
Irritability (General disorders) | 19 (20) | 33 (33)
Pyrexia (General disorders) | 160 (193) | 307 (364)
Jaundice (Hepatobiliary disorders) | 31 (31) | 45 (46)
Bronchiolitis (Infections and infestations) | 87 (98) | 132 (146)
Bronchitis (Infections and infestations) | 6 (8) | 19 (20)
Candida nappy rash (Infections and infestations) | 30 (30) | 52 (54)
Croup infectious (Infections and infestations) | 10 (10) | 27 (28)
Gastroenteritis (Infections and infestations) | 113 (128) | 196 (223)
Gastroenteritis viral (Infections and infestations) | 10 (12) | 22 (24)
Impetigo (Infections and infestations) | 9 (9) | 16 (17)
Lobar pneumonia (Infections and infestations) | 10 (11) | 14 (14)
Lower respiratory tract infection (Infections and infestations) | 53 (58) | 66 (70)
Nasopharyngitis (Infections and infestations) | 14 (14) | 38 (42)
Oral candidiasis (Infections and infestations) | 70 (75) | 118 (128)
Otitis externa (Infections and infestations) | 3 (3) | 19 (19)
Otitis media (Infections and infestations) | 268 (381) | 522 (742)
Otitis media acute (Infections and infestations) | 10 (10) | 17 (17)
Pneumonia (Infections and infestations) | 45 (50) | 97 (103)
Respiratory tract infection viral (Infections and infestations) | 17 (17) | 30 (32)
Skin candida (Infections and infestations) | 11 (11) | 20 (21)
Upper respiratory tract infection (Infections and infestations) | 459 (747) | 903 (1560)
Urinary tract infection (Infections and infestations) | 18 (18) | 22 (26)
Viral infection (Infections and infestations) | 80 (98) | 175 (217)
Viral skin infection (Infections and infestations) | 15 (15) | 31 (32)
Viral upper respiratory tract infection (Infections and infestations) | 32 (33) | 76 (78)
Cardiac murmur (Investigations) | 12 (12) | 35 (35)
Dehydration (Metabolism and nutrition disorders) | 10 (11) | 18 (18)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 18 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 65 (70) | 149 (171)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 55 (58) | 128 (140)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 47 (49) | 93 (104)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 71 (77) | 118 (123)
Dermatitis (Skin and subcutaneous tissue disorders) | 20 (21) | 39 (39)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 21 (23) | 24 (26)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 12 (12) | 18 (18)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 149 (183) | 298 (359)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (22) | 39 (40)
Eczema (Skin and subcutaneous tissue disorders) | 55 (62) | 80 (87)
Rash (Skin and subcutaneous tissue disorders) | 56 (61) | 135 (146)
Rash generalised (Skin and subcutaneous tissue disorders) | 3 (3) | 18 (18)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 18 (18) | 45 (47)
Flatulence (Gastrointestinal disorders) | 5 (5) | 15 (16)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 8 (8) | 8 (8)
Respiratory syncytial virus infection (Infections and infestations) | 10 (10) | 10 (10)
Rhinitis (Infections and infestations) | 8 (8) | 8 (8)
Heat rash (Skin and subcutaneous tissue disorders) | 4 (4) | 15 (16)
Seborrhoea (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it is understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.